CLINICAL TRIAL: NCT05933642
Title: Diuretic Efficacy of Aminophylline and Furosemide Combination vs Furosemide Alone in Critically Ill Adults
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Ng Haw Shyan, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202334-12198
Record Dates: First submitted 2023-06-14; First posted 2023-07-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Acute Kidney Injury
Keywords: Aminophylline; Furosemide; Critically ill; Adults; Intensive Care Unit (ICU)
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Aminophylline; Furosemide

STUDY DESIGN:
Intervention Model Description: double blind, randomised, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Recruited patient randomised into intervention vs control group by non clinical personnel, trial drugs dilution by research assistant, drug administered to patient by staff nurses, data collection by independent group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Intravenous (IV) infusion of (aminophylline 150mg and frusemide 120mg diluted to 50ml NS), IV load 10ml over 60 minutes, followed by IV infusion of 4 ml/hour
  Interventions: Drug: Aminophylline; Drug: Frusemide
- Control group (Active Comparator): IV infusions of furosemide (120mg diluted to 50ml NS), IV load 10ml over 60 minutes, followed by IV infusion of 4 ml/hour
  Interventions: Drug: Frusemide

INTERVENTIONS:
Drug: Aminophylline — aminophylline 150mg
  Arms: Treatment group
Drug: Frusemide — frusemide 120mg
  Other Names: Lasix

SUMMARY:
The goal of this RCT is to compare the effectiveness of aminophylline and furosemide combination vs furosemide alone in producing effective diuresis in critically ill adults in ICU. ICU patients with the need of improved diuresis will be recruited and given either infusion of aminophylline and furosemide combination or furosemide alone, and their hourly urine output will be monitored to compare their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and above who are admitted to the ICU of UMMC during the study period
* Oliguric patients, with the need for improved diuresis at clinician discretion - defined as urine output <0.5ml/kg/hour

Exclusion Criteria:

* Patient refusal for participation of study
* Patients with known hypersensitivity reaction to aminophylline or furosemide
* Patients with history of tachyarrhythmias, seizures, aspartate aminotransferase or alanine aminotransferase > 3 times normal, or hypothyroidism.

Patient with existing peptic ulcer disease or coagulopathy with INR > 1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-02 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with effective diuresis at 6 hours post intervention | 6 hours post intervention
  whether effective diuresis is achieved at 6 hours post intervention. Effective diuresis is defined as urine output >0.5ml/kg/hour based on patient's actual body weight

SECONDARY OUTCOMES:
Percentage of patients with effective diuresis at 2 hours post intervention | 2 hours post intervention
  whether effective diuresis is achieved at 2 hours post intervention. Effective diuresis is defined as urine output >0.5ml/kg/hour based on patient's actual body weight
Mean duration of infusion to achieve effective diuresis post intervention | Up to 6 hours post interventions
  Time in hours taken for infusion to achieve effective diuresis post intervention. Effective diuresis is defined as urine output >0.5ml/kg/hour based on patient's actual body weight
Changes in urine output at 6 hours post intervention | 6 hours post interventions
  Difference of hourly urine output (ml/hour) measured immediately before starting intervention and 6 hours post intervention
Changes in serum creatinine at 1 day post intervention | 1 day post intervention
  Difference of serum creatinine in mmol/l on the day of intervention and one day after intervention
Changes in serum eGFR at 1 day post intervention | 1 day post intervention
  Difference of serum eGFR in mL/min/1.73m2 on the day of intervention and one day after intervention
Percentage of patients requiring Renal Replacement Therapy (RRT) | throughout ICU stay, an average of 1 month
  Percentage of patients undergoing RRT during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Haw Shyan Ng, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No